CLINICAL TRIAL: NCT02194491
Title: A Phase 1 11β-Hydroxysteroid Dehydrogenase 1 Enzyme Occupancy Study Using a Positron Emission Tomography Ligand [11C]AS2471907- ([11C]MOZAT) and Following Single Oral Dose Administration of ASP3662 in Healthy Male Adult Subjects
Brief Title: A Positron Emission Tomography Occupancy Study Using Ligand [11C]AS2471907 and Following Oral Dosing of ASP3662
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3662-CL-0011
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Pharmacokinetics of ASP3662; Displacement of Radiotracer; Healthy Volunteers
Keywords: [11C]AS2471907; ASP3662; Positron Emission Tomography (PET); Brain enzyme occupancy
MeSH Terms: interventions — AS2471907; Magnetic Resonance Spectroscopy; ASP3662

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- [11C]AS2471907 administration (Part 1) (Experimental): Up to 4 single dose IV administrations (≤ 10 mL infused over approximately 1 minute) are planned, totaling less than 100 μg.
  Interventions: Other: [11C]AS2471907; Radiation: Positron Emission Tomography (PET)
- ASP3662 administration (Part 2) (Experimental): The dose levels used in part 2 will depend on the ongoing analysis of EO (enzyme occupancy) from previously dosed subjects.
  Interventions: Radiation: Positron Emission Tomography (PET); Drug: ASP3662

INTERVENTIONS:
Other: [11C]AS2471907 — intravenous radiotracer
  Other Names: Up to 4 single dose IV administrations (≤ 10 mL infused over approximately 1 minute) are planned; totaling less than 100 μg.
  Arms: [11C]AS2471907 administration (Part 1)
Radiation: Positron Emission Tomography (PET) — Imaging scanning procedure
Drug: ASP3662 — oral
  Arms: ASP3662 administration (Part 2)

SUMMARY:
The purpose of this study is to evaluate a novel PET tracer ([11C]AS2471907), and to use [11C]AS2471907 to assess the level and time-course of enzyme occupancy in the human brain prior to and following single oral dose administration of ASP3662.

DETAILED DESCRIPTION:
This is a two-part study where Part 1 will assess the test/retest variability of the ligand ([11C]AS2471907). Part 2 will assess the level and time-course of enzyme occupancy following ASP3662 dosing. Subjects will be confined to the clinic for up to 2 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject is of non-Asian descent.
* Subject has a body mass index (BMI) range of 18.5 to 32 kg/m2, inclusive and weighs at least 50 kg at screening.
* Subject and his female spouse/partner who is of childbearing potential must be using highly effective contraception1 consisting of 2 forms of birth control (at least one of which must be a barrier method) starting at screening and continuing throughout the study period and for 90 days after final study drug administration.
* Subject must not donate sperm starting at screening, throughout the study period and for at least 90 days after final study drug administration.
* Subject agrees not to participate in another investigational study while on study treatment.

Exclusion Criteria:

* Subject has a known or suspected hypersensitivity to ASP3662, [11C]AS2471907 or intolerance of drugs with the same mechanism of action as ASP3662.
* Subject has an allergy to topical anesthetics, such as, lidocaine (if used for catheter placement).
* Subject has previously participated in a clinical study with ASP3662 or part 1 of the current study.
* Subject has any of the liver enzymes (aspartate aminotransferase [AST], alanine transaminase [ALT], alkaline phosphatase [ALP], gamma-glutamyl transferase [GGT]) or total bilirubin (TBIL) above the upper limit of normal (ULN). If any liver enzyme is > 1 x ULN but ≤ 1.5 x ULN, the assessment may be repeated once during the screening period or on check-in. If the repeated assessment is above the ULN, it is exclusionary. If the initial value is > 1.5 x ULN, it cannot be repeated and is exclusionary.
* Subject has any clinically significant history of allergic conditions.
* Subject with a history of a suicide attempt or suicidal behavior.
* Subject has a history of smoking within the past 6 months.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal (GI), endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy, as judged by the investigator or designee.
* Subject has/had febrile illness or symptomatic viral, bacterial (including upper respiratory infection) or fungal (non-cutaneous) infection within 1 week before clinic check-in.
* Subject has any clinically significant abnormality following the investigator's review of the physical examination, electrocardiogram (ECG) and protocol-defined clinical laboratory tests at screening or clinic check-in.
* Subject has a mean pulse < 40 or > 90 beats per minute; mean systolic blood pressure > 140 mmHg or mean diastolic blood pressure > 90 mmHg (measurements taken in triplicate after subject has been resting in supine position for 10 minutes) at screening. If the mean pulse or mean systolic blood pressure (SBP) or mean diastolic blood pressure (DBP) is out of the range specified above, 1 additional triplicate measurement may be taken at screening.
* Subject has a mean QTcF interval of > 430 msec at screening or check-in. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken at screening. If this triplicate also gives an abnormal result, the subject should be excluded.
* Subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsade de pointes, structural heart disease or a family history of Long QT Syndrome.
* Subject has use of any prescribed or non-prescribed drugs (including vitamins, natural and herbal remedies, e.g., St. John's wort) in the 2 weeks before study drug administration, except for occasional use of acetaminophen (up to 2 g/day).
* Subject has history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical or substance abuse within the past 2 years prior to screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor) or the subject tests positive at screening or clinic admission for alcohol or drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates).
* Subject has any use of drugs of abuse within 3 months before screening or check-in.
* Subject has use of any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to check-in.
* Subject has consumed any caffeine-containing product within 24 hours prior to admission or grapefruit or star fruit within 7 days prior to admission.
* Subject has any significant blood loss, donated equal to 1 unit (450 mL) or more of blood or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days before check-in.
* Subject has a positive serology test for hepatitis B surface antigen, anti-hepatitis A virus (Immunoglobulin M), anti-hepatitis C virus or anti-human immunodeficiency virus (HIV) Type 1 or Type 2 at screening.
* Subject has participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half-lives, whichever is longer, before the initiation of screening.
* Subject is an employee of the Astellas Group or vendors involved in the study.
* Additionally, a subject who meets the following imaging exclusion criteria will not be included in this study:

  * Subject who suffers from claustrophobia.
  * Subject who has received a diagnostic or therapeutic radiopharmaceutical within 7 days prior to participation in this study.
  * Participation in other research studies involving ionizing radiation within 1 year of the PET scans that would cause the subject to exceed the US Nuclear Regulatory Commission yearly dose limits for healthy subjects, i.e., an effective dose of 5 Roentgen equivalent man (rem) received per year.
  * Subject with history of IV drug use which would prevent venous access for PET tracer injection.
  * Severe motor problems that prevent the subject from lying still for PET imaging.
  * Subject who has chronic pain for any reason (e.g., as the result of rheumatoid arthritis).
  * Subject who has an MRI scan deemed to be structurally abnormal by the investigator and thus precluding proper identification of the regions of interest (ROIs) (e.g., cortical atrophy). The MRI scan for an individual subject may be omitted if the required anatomical MRI scan for this subject is on file and was performed within approximately 6 months prior to dosing, as part of participation in an approved Yale Protocol.
  * Subjects who has current, past or anticipated exposure to radiation in the work place.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Positron Emission Tomography measure: volume of distribution | Day 1 and 2 (Part 1 and Part 2)
Positron Emission Tomography measure: brain time-activity curves | Day 1 and 2 (Part 1 and Part 2)
Positron Emission Tomography measure: enzyme occupancy | Day 1 and 2 (Part 1 and Part 2)
Positron Emission Tomography measure: binding potentials | Day 1 and 2 (Part 1 and Part 2)
Pharmacokinetic parameter of ASP3662 and its metabolite (AS2570469): AUClast (Part 2 only) | Day 1 and 2
  Area under the plasma concentration - time curve from time zero to time of last measurable concentration (AUClast)
Pharmacokinetic parameter of ASP3662 and its metabolite (AS2570469): Cmax (Part 2 only) | Day 1 and 2
  Maximum concentration (Cmax)
Pharmacokinetic parameter of ASP3662 and its metabolite (AS2570469): tmax (Part 2 only) | Day 1 and 2
  Time to attain Cmax (tmax)
Safety as assessed by laboratory tests, 12-lead electrocardiograms, vital signs, adverse events, physical exams, neurological exams and Columbia Suicide Severity Rating Scale | up to 9 days (Part 1 and Part 2)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Site US10001, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided